CLINICAL TRIAL: NCT06204887
Title: Evaluation of Different Irrigation-Activation Techniques on Healing Outcome of Large Periapical Lesions: A Randomized Controlled Trial
Brief Title: Effect of Irrigation-Activation Techniques on Healing in Large Periapical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Ahter Sanal Cikman, Assistant Professor, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/35
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Effect of Irrigation Activation on Periapical Healing
Keywords: Irrigation activation; periapical healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Manual dynamic activation (Experimental)
  Interventions: Procedure: Manual dynamic activation
- Passive ultrasonic activation (Experimental)
  Interventions: Procedure: Passive ultrasonic activation
- Laser activation (Experimental)
  Interventions: Procedure: Laser activation
- Non-activated Control (No Intervention)

INTERVENTIONS:
Procedure: Manual dynamic activation — The root canals were filled with irrigation solutions. A main gutta percha cone was positioned 1 mm shorter than the working length and 2 mm coronal-apical direction movement was performed at a rate of 100 strokes per minute during 60 s.
  Arms: Manual dynamic activation
Procedure: Passive ultrasonic activation — A non-cutting ultrasonic tip (IRRI S 21/25; VDW, Munich, Germany) coupled to an ultrasonic device (DTE S6 Led, Guilin Woodpecker Co., Guilin, Guangxi, China) (mode: E, setting: 6) was used according to the manufacturer's recommendations.
  Arms: Passive ultrasonic activation
Procedure: Laser activation — A 2940 nm Er:YAG-laser device (Lightwalker, Fotona, Ljubljana, Slovenia), equipped with a handpiece (H14, Fotona) holding a 8.5 mm long and 600 µm diameter-tapered fiber tip (SWEEPS 600, Fotona) was used for irrigation activation. The device was set to AutoSWEEPS mode with two ultrashort micropulse durations (25 μs) continuously varying at 0.3 W, 20 mJ, 15 Hz settings. The air and water sprays were turned off.
  Arms: Laser activation

SUMMARY:
The aim of this study was to highlight the healing rates of large periapical lesions after different irrigation activation treatments as manual dynamic activation (MDA), passive ultrasonic irrigation (PUI), shock wave-enhanced emission photoacoustic streaming (SWEEPS) using CBCT scans based on volumetric change analysis during 1-year follow-up.

DETAILED DESCRIPTION:
The aim of this study was to highlight the healing rates of large periapical lesions after different irrigation activation treatments as manual dynamic activation (MDA), passive ultrasonic irrigation (PUI), shock wave-enhanced emission photoacoustic streaming (SWEEPS) using CBCT scans based on volumetric change analysis during 1-year follow-up.

A total of 56 systemically healthy male/female patients with mandibular single-rooted teeth with a periapical index score (PAI) of 3 or higher were included in the study. Pretreatment lesion volumes were determined by CBCT. Patients were randomly divided into 3 study groups (PUI, SWEEPS, MDA) and control group (n=14). For the follow-up routine, 2D radiographs were taken at months 3, 6, and 9, as well as clinical examinations. At the end of 12 months, 3D evaluation of lesion volumes was performed using ITK SNAP. Pretreatment and follow-up values were statistically analyzed with the Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

* Patients having single root mandibular teeth
* Patients the diagnosis of chronic apical periodontitis,
* Periapical index score of 3 and above,
* Patients having good oral hygiene

Exclusion Criteria:

* Patients with systemic diseases (diabetes, hypertension, chronic liver disease, coagulation disorders),
* Patients with bone metabolism disease and/or
* Patients using drugs that affect bone metabolism (such as steroids, bisphosphonates)
* Patients with a history of radiotherapy
* Pregnant patients
* Teeth with mobility of 2 or more, periodontal pocket depth of 5 mm or more, generalized chronic periodontitis, internal and external resorption, and/or vertical and horizontal root fractures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahter Şanal Çıkman, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 97 enrolled participants, 70 met inclusion criteria and randomized to irrrigation protocols.
Groups:
- Non-activated Control: No activation protocol was applied during irrigation.
Period: Overall Study
Arm/Group | Manual Dynamic Activation | Passive Ultrasonic Activation | Laser Activation | Non-activated Control
Started | 17 | 18 | 15 | 20
Completed | 14 | 14 | 14 | 14
Not Completed | 3 | 4 | 1 | 6
Not completed — Lost to Follow-up | 3 | 4 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Dynamic Activation | Passive Ultrasonic Activation | Laser Activation | Non-activated Control | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 56
Age, Continuous [Mean (Full Range); unit: Years] | 34.071 [18 to 60] | 38 [20 to 64] | 41.928 [21 to 63] | 37.073 [21 to 58] | 37.768 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 8 | 4 | 22
  Male | 9 | 9 | 6 | 10 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 14 | 14 | 14 | 14 | 56
Pre-operative lesion volumes [Mean (Standard Deviation); unit: mm3] | 193.936 (29.441) | 158.343 (40.275) | 168.371 (37.904) | 172.2 (41.707) | 173.212 (37.331)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Lesion Volume at 12-months Follow-up
Description: 3D volumes pre-operatively and at the end of 1 year were measured using the segmentation technique by slicing the image at 0.09 mm intervals. The borders of the lesion were determined with gray scale. The defined volume boundaries were automatically filled by bubbles until the entire defect was filled completely. If necessary, manual correction was applied at this stage of lesion volume measurements, allowing for small individual additions or subtractions. At the end, the well-defined size of the lesion could be visualized in 3D. After finishing the process, the software depicted the exact volume of the defects in mm3.The volume data were compared with the preoperative CBCT measurements in each case. The primary healing of the periapical tissues was assessed, volume changes were measured, and the long-term outcomes of the procedures were compared using percentage of the lesion volume change.
Time Frame: One year from the beginning of the study
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Manual dynamic activation | Passive ultrasonic activation | Laser activation | Non-activated Control
Number analyzed (Participants) | 14 | 14 | 14 | 14
percent change | 80.429 (28.294) | 85.429 (8.635) | 86.929 (23.332) | 74.571 (36.515)
Statistical Analysis 1: Comparison: Manual dynamic activation vs Passive ultrasonic activation vs Laser activation vs Non-activated Control; Test type: Superiority; p < 0.05, Kruskal-Wallis

2. Primary Outcome: Distribution of Lesion Status in Different Irrigation Groups at 12-year Follow-up
Time Frame: One year from the beginning of the study
Measure: Number; unit: participant
Arm/Group | Manual dynamic activation | Passive ultrasonic activation | Laser activation | Non-activated Control
Number analyzed (Participants) | 14 | 14 | 14 | 14
participant
  Totally healed | 3 | 1 | 4 | 3
  Reduced | 9 | 13 | 9 | 8
  Unchanged | 2 | 0 | 1 | 3
  Enlarged | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Death, serious adverse events, and other(non-serious adverse events) were not assessed for the study.
Arm/Group | Manual Dynamic Activation | Passive Ultrasonic Activation | Laser Activation | Non-activated Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The follow-up period of the study was 1 year, which may have limited our ability to obtain definitive evidence of lesion changes in the long term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT06204887/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT06204887/SAP_001.pdf
  • Informed Consent Form (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT06204887/ICF_002.pdf